CLINICAL TRIAL: NCT06302686
Title: engAGE: Managing cognitivE decliNe throuGh Theatre Therapy, Artificial Intelligence and Social Robots drivEn Interventions
Acronym: engAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: INRCA_004_2023
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-04

CONDITIONS: Mild Cognitive Impairment; Older Adults
Keywords: ageing; older adults; mild cognitive impairment; caregiver; technological platform
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- engAGE group (Experimental): The experimental group will use the technological engAGE system for 6 months.
  Interventions: Device: engAGE system
- control group (Other): To the control group will be given a booklet containing information and activities on well-being to do at home.
  Interventions: Other: Group practicing with only the support of a booklet

INTERVENTIONS:
Device: engAGE system — The experimental group use the engAGE system at both healthcare organization and home. At the healthcare organization, the subject interacts with Pepper robot. The interaction is supervised by the formal caregivers and includes the following activities: dialoguing with the robot, storytelling, drama play, cognitive and physical games. This interaction is planned to last about 1 hour twice a week for 6 months. At home, the older user interacts with the tablet supervised by the informal caregiver. The user plays cognitive and physical games installed on MEMAS app. This activity is performed for 0.5 hour, every day for 6 months. Throughout the whole period of experimentation, the older user wears the smartwatch that measures his/her physiological parameters and the steps. Any activity performed by the seniors is assigned by formal caregiver and can be personalized taking into account the user's abilities, lifestyle, and social interactions.
  Arms: engAGE group
Other: Group practicing with only the support of a booklet — To the control group will be given a booklet containing information and activities on well-being to do at home.
  Arms: control group

SUMMARY:
The objectives of the engAGE project are to counteract and slow down cognitive decline progression, to enhance the intrinsic capacity of the users, and to support the wellbeing of older persons with mild cognitive impairment (MCI) by providing an ecosystem of services based on an innovative system that integrates social robots.

DETAILED DESCRIPTION:
The study is focused on older people with mild cognitive impairment, aiming to improve their quality of life and well-being, allowing them to preserve their identity, to reduce stress, memory loss, or communication challenges by the use of the technological engAGE system that includes the social robot Pepper. The social robot can be a great tool in engaging older adults in this kind of activities. It is always available and able to provide verbal clues or suggestions according to older adult's wishes, needs and memories. Moreover, the social robots may coach the older adults to perform daily activities with greater independence (i.e. coaching stepwise prompting to complete activities in-home) and support to caregivers as well.

Since caring for people with mild cognitive impairment puts a significant burden on informal caregivers, having the support of a technological platform can reduce anxiety, worries, and stress. The caregivers can personalize the content of interventions to the wishes and preferences of the older adults. Together with the older adults, they can be involved with the robot in joyful and fun activities like drama playing, storytelling, etc.

The formal caregivers who need to keep track of older adult progress which is a difficult and time-consuming process due to the lack of objective monitoring of cognitive decline and wellbeing may get valuable support from the cognitive assessment procedure implemented by the machine learning algorithm. Also, the social robot and tablet may facilitate the follow-up of older adults through reminders and cognitive interventions.

ELIGIBILITY:
Inclusion Criteria:

* mild cognitive impairment (MCI);
* Montreal Cognitive Assessment (MoCA) score 21 - 25;
* Memory Assessment Clinics - Questionnaire (MAC-Q) ≥ 25;
* Reisberg scale 2 - 4;
* Clinical Frailty Scale score 1 - 3;
* 4-items GDS score ≤ 1;
* have an informal caregiver to support in carrying out the main daily activities.

Exclusion Criteria:

* lack of informal caregivers;
* significant visual or hearing impairment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-06-24 (Estimated); Study Completion 2024-06-24 (Estimated)

PRIMARY OUTCOMES:
Change in perceived stability of cognitive status by the older adults | baseline and 6 months later
  The Memory Assessment Clinics - Questionnaire (MAC-Q) is a 6-item scale that uses a 5-item Likert scale from "much better now"=1 to "much worse now"=5, and the last question scores double. The questionnaire asks the person to compare his or her memory with a previous period to measure age-related memory decline. Five items address specific situations frequently reported as problematic by those who experience memory loss with age. One item is a global item assessing general memory decline. A cutoff of 25 points or more indicates that the individual has a memory disorder.

SECONDARY OUTCOMES:
Change in cognitive impairment in older adults | baseline and 6 months later
  The Montreal Cognitive Assessment (MoCA) is a screening assessment for detecting cognitive impairment. The MoCA assesses several cognitive domains: the short-term memory recall task (5 points), visuospatial abilities (4 points), alternation task (1 point), verbal abstraction task (1 point), attention, concentration, and working memory (6 points), language (6 points), abstract reasoning (2 points), and orientation to time and place (6 points).Scores on the MoCA range from zero to 30. A score of 26 and higher is considered normal.
Change in depression in older adults | baseline and 6 months later
  The 4-items Geriatric Depression Scale (GDS) is a 4-items scale whose answers are yes or no. If all the items are answered negatively then the depression is excluded; if only one item is answered positively then the situation is uncertain; if at least 2 items are answered positively, the patient is depressed.
Change in frailty status in older adults | baseline and 6 months later
  The Clinical Frailty Scale (CFS) is a descriptive scale divides the older participants into 9 classes based on the information provided by them and their relatives: between 1 and 3 the patient is non-frail, pre-frail if 4, he is frail from 5 to 9.
Change in mental well being in older adults | baseline and 6 months later
  The Warwick-Edinburgh Mental Wellbeing Scales (WEMWBS). is used to enable the measuring of mental wellbeing in the general population. The 12-item scale WEMWBS has 5 response categories, summed to provide a single score. Scores range from 7 to 35 and higher scores indicate higher positive mental wellbeing.
Change in quality of life in older adults | baseline and 6 months later
  The EuroQoL-5D-5L scale consists of five dimensions: mobility, independence, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, mild problems, moderate problems, severe problems and extreme problems. The numbers from the five dimensions can be combined into a 5-digit number that describes the health status of the participant.
Change in acceptability of the engAGE system in older adults | baseline and 6 months later
  Acceptability will be assessed by the Unified Theory of Acceptance and Use of Technology test (UTAUT). It's a standardized instrument for measuring the likelihood of success for new technology introductions and helps to understand the drivers of its acceptance.
  The questionnaire has 52 questions distributed in 4 key constructs: 1) performance expectancy, 2) effort expectancy, 3) social influence, and 4) facilitating conditions.
  Each question are based on a Likert-type 5-point scale ranging from 1 = strongly disagree to 5 = strongly agree. Increments are integers between 1 to 5.
Change in quality of life in informal caregivers | baseline and 6 months later
  The EuroQoL-5D-5L scale consists of five dimensions: mobility, independence, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, mild problems, moderate problems, severe problems and extreme problems. The numbers from the five dimensions can be combined into a 5-digit number that describes the health status of the participant.
Change in mental well being in informal caregivers | baseline and 6 months later
  The Warwick-Edinburgh Mental Wellbeing Scales (WEMWBS) is used to enable the measuring of mental wellbeing in the general population. The 12-item scale WEMWBS has 5 response categories, summed to provide a single score. Scores range from 7 to 35 and higher scores indicate higher positive mental wellbeing.
Change in caregiver burden | baseline and 6 months later
  The Zarit Burden Interview (ZBI) is a caregiver self-report measure, containing 22 items. Each item on the interview is a statement which the caregiver is asked to endorse using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always).

CONTACTS AND LOCATIONS:
Locations (3):
- IRCCS INRCA Hospital, Ancona, Italy
- Karde A/S, Oslo, Norway
- HUG, Geneva, Switzerland

REFERENCES:
- [Derived] Amabili G, Maranesi E, Margaritini A, Bonfigli AR, Felici E, Barbarossa F, Benadduci M, Gosetto L, Guebey J, Grimstad T, Hellman R, Marin AI, Boye LT, Anghel IM, Cioara T, Bevilacqua R. Managing Cognitive Decline Through a Social Robot-Based Intervention: Protocol for the engAGE Proof of Concept and Randomized Controlled Trial. JMIR Res Protoc. 2025 Sep 2;14:e67601. doi: 10.2196/67601. PMID 40896828